CLINICAL TRIAL: NCT06638918
Title: Assessing the Feasibility of a Virtual Reality Intervention for Lower Phantom Limb Pain in the Acute Postoperative Period
Brief Title: Assessing the Feasibility of a Virtual Reality Intervention for Phantom Pain Immediately Following Lower Limb Amputation
Status: Completed | Type: Observational
Sponsor: University of Manitoba (Other)
Collaborators: Health Sciences Centre, Winnipeg, Manitoba (Other)
Responsible Party: Principal Investigator, Renée El-Gabalawy, Associate Professor & Clinical Psychologist, University of Manitoba
Other Study IDs: HS25778
Record Dates: First submitted 2024-09-04; First posted 2024-10-15 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Phantom Limb Pain
Keywords: virtual reality; phantom limb pain; lower limb amputation; graded motor imagery; feasibility; acute
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Virtual Reality Group: These participants will receive the virtual reality intervention for at least 20 minutes daily for approximately seventeen sessions, or as long as they are able.
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Device: Virtual Reality — The virtual reality (VR) intervention administers graded motor imagery (GMI) treatment for phantom limb pain. It consists of three stages: left right sorting task (a sorting task where participants sort images of left and right feet), explicit motor imagery (a series of guided imagery exercises administered via audio to facilitate focus on the phantom limb), and the limb simulation task (where participants perform a series of exercises with virtual legs to create the illusion of movement in their phantom limb). The limb simulation stage can also be conducted with leg trackers to generate a higher degree of illusion in the virtual legs.

SUMMARY:
The goal of this observational study is to see whether a new virtual reality (VR) program meant to treat phantom limb pain (PLP) is feasible to people immediately following lower limb amputation. This study aims to answer three questions.

1. Is this VR treatment acceptable to people immediately following lower limb amputation?
2. Are the researchers able to recruit participants that represent the population in need of this treatment, and will these participants stay until the end of the study?
3. Do participants who use the VR program more have less severe PLP than participants who use the VR program for fewer sessions?

Participants will:

* Try the VR program in the hospital, their home, and in physiotherapist clinics daily for about seventeen sessions.
* After each session, participants will fill out questionnaires asking about their level of pain, their nausea, and how acceptable they find the program. They will also complete measures asking about how they're feeling and what led to their amputation.
* One month following their final VR session, researchers will phone the participants to ask them to rate how severe their PLP is.

DETAILED DESCRIPTION:
There are many barriers that prevent people with lower limb amputations (LLA) from receiving effective nonpharmacological treatment for their phantom limb pain (PLP), such as long outpatient wait times and the sparse number of amputation rehabilitation specialists. Early administration of effective PLP treatments, such as graded motor imagery (GMI), may improve both treatment access and efficacy if it is administered through virtual reality (VR). However, no VR GMI treatments have been developed or tested in the acute postoperative period following LLA to prevent PLP. The current study will recruit 30 patients being treated for LLA at the Health Sciences Centre (HSC) in Winnipeg, Manitoba to assess the feasibility and pilot outcomes of a novel VR GMI program administered in the postoperative acute care setting, with the goal of preventing and or reducing PLP. First, the researchers predict the mean acceptability, tolerability, and length of engagement in the VR program will be high across administration contexts and each of the VR stages. Second, the researchers hypothesize the recruitment strategies employed will capture and retain a large, representative sample of individuals undergoing LLA at the HSC. Lastly, the researchers predict length of VR program engagement will demonstrate a preliminary effect on PLP incidence, intensity, and interference at one-month follow-up. Baseline characteristics such as anxiety, depression, and amputation etiology will also be explored as extraneous variables. This research will be the first to provide evidence for the feasibility of VR PLP treatment administered immediately following LLA. The results will inform future development of the VR program and optimize the study procedures for an upcoming randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* if they underwent or are about to undergo an LLA (hip, below-knee, above-knee, or foot) within the last two months
* if they are currently receiving inpatient treatment at the Health Sciences Centre (HSC) in Winnipeg, Canada
* if they can speak/read English fluently

Exclusion Criteria:

* any visual, hearing, or motor impairment that would affect engaging with a head-mounted VR headset or hand controls, as interpreted by the research team or nursing staff

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from population of individuals undergoing lower limb amputation at the Health Sciences Center (a public inpatient tertiary care hospital) in Winnipeg, Manitoba.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-07-26 (Actual); Primary Completion 2025-10-17 (Actual); Study Completion 2026-01-05 (Actual)

PRIMARY OUTCOMES:
Acceptability | Immediately after intervention is administered
  The Theoretical Framework of Acceptability Questionnaire (TFAQ score > 3 indicates acceptability). Range 1-5 on seven items.
Tolerability of the virtual reality simulation | Immediately before and after intervention administration
  Numerical Rating Scale for phantom limb pain, residual limb pain (i.e., physical pain at the amputation site), nausea (NRS > 2 on any construct indicates an adverse event and lack of tolerability). Range 0-10 on each NRS.
Engagement | During intervention administration, up to seventeen days
  Length of time in minutes spent in the virtual reality program per session (recommended: 20 minutes)

SECONDARY OUTCOMES:
Phantom Limb Pain Intensity | One month follow-up
  Brief Pain Inventory (Pain Intensity Only). Range 0-40, higher scores = higher pain intensity.
Phantom Limb Pain Interference | One month follow-up
  Patient-Reported Outcome Measurement System Pain Interference Scale-- 8a. Range 8-40, higher score = higher pain interference.
Embodiment | Administered after intervention administration is completed, up to seventeen days
  Virtual Embodiment Questionnaire. Range 1-7 for 12 items, higher score = higher embodiment.
Presence | Administered after intervention administration is completed, up to seventeen days
  iGroup Presence Questionnaire. Range -3 to +3 for each of 14 items, higher score = higher presence.

OTHER OUTCOMES:
Anxiety | Baseline
  Generalized Anxiety Disorder 7. Range 0 to 21, higher score = higher anxiety.
Depression | Baseline
  Patient Health Questionnaire 9. Range 0 to 27, higher score = higher depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Renee El-Gabalawy, PhD, Principal Investigator — Associate Professor and Clinical Psychologist
Locations (1):
- Health Sciences Center, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No
It is not typical to share the individual participant data from a feasibility study.

REFERENCES:
- [Derived] El-Gabalawy R, Crooks M, Smith MSD, Hammond E, Gross P, Roznik M, Perrin D, Reynolds K, Logan G, Pankratz L, Johnson H, Girling L, Wiebe D. Treating Lower Phantom Limb Pain in the Postoperative Acute Care Setting Using Virtual Reality: Protocol for a 4-Phase Development and Feasibility Trial. JMIR Res Protoc. 2025 May 23;14:e68008. doi: 10.2196/68008. PMID 40409745